CLINICAL TRIAL: NCT00698594
Title: Comparison of Effectiveness and Safety of Sublingual Immunotherapy in Children With Allergic Rhinitis Allergic to Grass Pollen
Brief Title: Comparison of Effectiveness and Safety of Sublingual Immunotherapy in Children With Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, Head of the Department of Pediatrics and Allergy, Medical University of Lodz, N. Copernicus Hospital, MD, PhD, Prof., Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RNN/98/08/KE
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Group of children with allergic rhinitis 6-18 years old. receiving seasonally grass pollens sublingual allergen extract (Staloral 300 IR, Stallergenes, France) (n=20) - seasonal SLIT group
  Interventions: Biological: sublingual allergen extract
- 2 (Active Comparator): Group of children with allergic rhinitis 6-18 years old receiving yearly grass pollens sublingual allergen extract (Staloral 300 IR, Stallergenes, France) (n=20) - yearly SLIT group
  Interventions: Biological: sublingual allergen extract
- 3 (Placebo Comparator): Group of children with allergic rhinitis 6-18 years old receiving placebo in sublingual applicator (Staloral 300 IR, Stallergenes, France) (n=20) - placebo group
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: sublingual allergen extract — Group of children with allergic rhinitis 6-18 years old. receiving seasonally grass pollens sublingual allergen extract (Staloral 300 IR, Stallergenes, France) (n=20) - seasonal SLIT group
  Other Names: Staloral 300 IR, Stallergenes, France
  Arms: 1
Biological: sublingual allergen extract — Group of children with allergic rhinitis 6-18 years old receiving yearly grass pollens sublingual allergen extract (Staloral 300 IR, Stallergenes, France) (n=20) - yearly SLIT group
  Other Names: Staloral 300 IR, Stallergenes, France
  Arms: 2
Biological: placebo — Group of children with allergic rhinitis 6-18 years old receiving placebo in sublingual applicator (Staloral 300 IR, Stallergenes, France) (n=20) - placebo group
  Arms: 3

SUMMARY:
The purpose of the trial is to compare the efficacy and safety of sublingual seasonal and annual immunotherapy in children with allergic rhinitis allergic to grass pollens.

DETAILED DESCRIPTION:
Allergen immunotherapy is currently the only one method of cause treatment of the IgE-dependent allergic diseases. Sublingual immunotherapy (SLIT) is the method which allows to give allergens via alternative oral route in patients home. Due to the possibility of avoiding injection this therapy allows to have better relationship with patient, and reduce the costs of therapy thanks to reducing the numbers of visits in out-patient clinic.However efficacy and safety of sublingual immunotherapy are still important issues, especially in children.

The purpose of trial is to compare the efficacy and safety of sublingual seasonal and annual immunotherapy in children with allergic rhinitis allergic to grass pollens.

ELIGIBILITY:
Inclusion Criteria:

* Children with seasonal allergic rhinitis, allergic to grass pollens, first diagnosed at least 2 years before inclusion into the study

Exclusion Criteria:

* Active upper respiratory tract infection within 3 weeks before the study and acute sinus disease requiring antibiotic treatment within 1 month before the study
* Allergic rhinitis hospitalisation during the 3 months before the first visit.
* Additional criteria were other clinically significant pulmonary, hematologic, hepatic, gastrointestinal, renal, endocrine, neurologic, cardiovascular, and/or psychiatric diseases or malignancy that either put the patient at risk when participating in the study or could influence the results of the study or the patient's ability to participate in the study as judged by the investigator.
* Excluded medications were systemic corticosteroids.
* Patients who were receiving immunotherapy were also excluded.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Clinical symptoms of allergic rhinitis (Pediatric Quality of Life Questionnaire) | Following visits after starting the study: at 6 months, 9 months, 12 months, 18 months, 21 months, 24 months.
  Visit 2 (6 months after starting the study), visit 3 (9 months after starting the study), visit 4 (12 months after starting the study), visit 5 (18 months after starting the study), visit 6 (21 months after starting the study), visit 7 (24 months after starting the study).

SECONDARY OUTCOMES:
Change of percent of regulatory lymphocytes in the peripheral blood. | at baseline and at the end of the second season (22 months interval)
non-specific bronchial hyperreactivity with methacholine (PC20M), specific nasal provocation test. | at the end of the first and second season of the study (12 months interval)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Stelmach, Prof., Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Poland, Lodz, Łódź Voivodeship, Poland